CLINICAL TRIAL: NCT00503412
Title: A Phase 1, Open Label, Non-Randomised, Single Centre Pharmacokinetic and Mass Balance Study of Orally Administered 14-C-AZD2171 in Patients With Solid Metastatic Tumours
Brief Title: Phase I Orally Administered 14C-AZD2171 in Patients With Solid Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00019
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Solid Metastatic Tumor
Keywords: phase I; AZD2171; solid tumor; metastatic tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD2171 — oral 14C
  Other Names: cediranib; RECENTIN™

SUMMARY:
Open, non-randomised, radiolabelled, single centre study with a total of six patients with solid metastatic tumors to determine the rates and routes of elimination of 14C-AZD2171 and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastatic tumor which is refractory to standard therapies
* life expectancy is 12 weeks or longer
* WHO performance status is 0-12

Exclusion Criteria:

* radiotherapy and chemotherapy within 4 weeks before the start of the study treatment
* patients with a history of poorly controlled hypertension
* history or evidence of any medical condition that might affect gastrointestinal function
* patients that have participated in a radiolabelled study in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the rates & routes of excretion of 14C radiolabelled AZD2171 in patients by assessment of concentrations of total 14C radioactivity and AZD2171 in plasma & concentrations of total radioactivity in urine&faeces | assessed at time intervals post dose

CONTACTS AND LOCATIONS:
Overall Officials: Nick Botwood, BSc, MBBS, MRCP, MFPM, Study Director — AstraZeneca; Stan Kaye, Prod, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Research Site, Sutton, United Kingdom